CLINICAL TRIAL: NCT05924412
Title: A Randomized Comparison Between Parecoxib and Placebo Added to a Standard Perioperative Analgesic Protocol for Total Knee Arthroplasty
Brief Title: Parecoxib in Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Julian Aliste, Associate Professor, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OAIC1308/22
Record Dates: First submitted 2023-06-08; First posted 2023-06-29 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Pain, Postoperative; Pain, Acute; Analgesia; Analgesic Nephropathy; Analgesic Adverse Reaction; Knee Osteoarthritis
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Agnosia; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parecoxib (Experimental): This arm will receive intravenous parecoxib in the intraoperative period.
  Interventions: Drug: Intravenous study drug
- Placebo (Placebo Comparator): This arm will receive a placebo intravenous injection containing saline solution in the same volume as the intervention group
  Interventions: Other: Intravenous saline solution

INTERVENTIONS:
Drug: Intravenous study drug — 40mg parecoxib will be administered intravenously after general anesthesia induction and before tourniquet inflation and surgical incisión
  Arms: Parecoxib
Other: Intravenous saline solution — Saline solution (same volume as the study drug) will be administered intravenously after general anesthesia induction and before tourniquet inflation and surgical incision
  Arms: Placebo

SUMMARY:
Early mobilization and rehabilitation can be difficult after total knee arthroplasty (TKA) due to a high incidence of moderate to severe postoperative pain. Non-steroidal anti-inflammatory drugs (NSAIDs) are important to multimodal analgesic protocols. Parecoxib is an NSAID that selectively inhibits the enzyme cyclooxygenase-2 (COX-2). Clinical trials have shown that it does not alter platelet function or gastric mucosa. A recent study, after comparing ketorolac and parecoxib used at the same time in infiltration and systemically, found no differences in perioperative analgesia with a tendency to less bleeding in the parecoxib group. This randomized study will compare the effectiveness of adding a COX-2 inhibitor in the pain management of patients undergoing TKA as part of a multimodal analgesia regimen. The morphine consumption was selected as the primary outcome. The study hypothesis is that patients receiving parecoxib would have a lower opioid consumption.

ELIGIBILITY:
Inclusion Criteria:

ASA I - III BMI 20 - 35 (kg/m2)

Exclusion Criteria:

* Adults who are not capable of giving their own consent
* Pre-existing neuropathy (assessed in the history and physical examination)
* Coagulation disturbance (assessed on history and physical examination, if clinically necessary, by blood test, i.e. platelets ≤ 100,000, international normalized ratio ≥ 1.4 or prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination, if considered clinically necessary, by blood test, i.e. creatinine ≥ 1.04 mg/dl)
* Hepatic impairment (assessed by history and physical examination, if considered clinically necessary, by blood tests, i.e. transaminases (GGT ≥ 50 u/lt)
* Allergy to local anesthetics, morphine, paracetamol, ketorolac or parecoxib
* Pregnancy
* Chronic pain syndromes that require the use of opioids at home
* Known history of sulfa allergy
* History of ischemic heart disease
* History of chronic gastritis or peptic ulcer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours
  Morphine consumed postoperatively during the first 24 hrs utilizing a patient-controlled analgesia device programmed 1mg/ml morphine solution, no infusion, 1ml dose, 8 minutes lockout.

SECONDARY OUTCOMES:
Basal quadriceps strength in the operative side | 1 hour before surgery
  Leg extension strength measured with a handheld dynamometer
Basal level of pain during leg extension in the operative side | 1 hour before surgery
  Pain level measured with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Basal plasmatic creatinine | 1 hour before surgery
  Plasmatic creatinine level measured in mg/dL from a blood sample
Nerve block performance time | 5 minutes after anesthesia induction (before surgical incision)
  Time elapsed between skin disinfection and the end of local anesthetic injection in femoral triangle and posterior capsule blocks.
Incidence of Block complications | 5 minutes after anesthesia induction and before surgical incision
  Report of vascular puncture, hematoma, local anesthetic systemic toxicity symptoms
Time to first morphine dose request | 24 hours
  Time in minutes between arrival to post anesthesia care unit arrival and first request of morphine with the patient controlled analgesia device
Morphine consumption during first 48 hours | 48 hours
  Morphine consumed postoperatively during the first 48 hrs utilizing a patient-controlled analgesia device programmed 0.01mg/Kg/ml morphine solution, no infusion, 1ml dose, 8 minutes lockout.
Incidence of opioid related side effects | 48 hours
  Report of nausea, vomitus, pruritus, urinary retention, respiratory depression
Incidence of NSAIDs related clinical side effects | 48 hours
  Report of allergic reactions, pyrosis, evident gastrointestinal bleeding, hematoma
Postoperative static pain level at 3 hours | 3 hours
  Pain level measured at rest with an 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative dynamic pain level at 3 hours | 3 hours
  Pain level measured during leg extension with an 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative static pain level at 6 hours | 6 hours
  Pain level measured at rest with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative dynamic pain level at 6 hours | 6 hours
  Pain level measured during leg extension with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative static pain level at 12 hours | 12 hours
  Pain level measured at rest with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative dynamic pain level at 12 hours | 12 hours
  Pain level measured during leg extension with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative static pain level at 24 hours | 24 hours
  Pain level measured at rest with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative dynamic pain level at 24 hours | 24 hours
  Pain level measured during leg extension with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative static pain level at 48 hours | 48 hours
  Pain level measured at rest with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Postoperative dynamic pain level at 48 hours | 48 hours
  Pain level measured during leg extension with a 11-points numeric rating scale (from 0 to 10 where 0 means absence of pain and 10 the worst imaginable pain)
Medial malleolus sensory block level | 3 hours
  0 to 2 points for Sensory block to cold and touch in the medial malleolus. 0 point= can feel cold and touch; 1= can feel touch but not cold; 2= cannot feel cold or touch
Lateral malleolus sensory block level | 3hours
  0 to 2 points for Sensory block to cold and touch in the medial malleolus. 0 point= can feel cold and touch; 1= can feel touch but not cold; 2= cannot feel cold or touch
Medial malleolus sensory block level | 24 hours
  0 to 2 points for Sensory block to cold and touch in the medial malleolus. 0 point= can feel cold and touch; 1= can feel touch but not cold; 2= cannot feel cold or touch
Lateral malleolus sensory block level | 24 hours
  0 to 2 points for Sensory block to cold and touch in the medial malleolus. 0 point= can feel cold and touch; 1= can feel touch but not cold; 2= cannot feel cold or touch
Postoperative quadriceps strength | 3 hours
  Leg extension strength measured with a handheld dynamometer
Postoperative quadriceps strength | 24 hours
  Leg extension strength measured with a handheld dynamometer
Incidence of restriction to perform physiotherapy | 6 hours
  Inability to perform physiotherapy secondary to pain or motor blockade
Incidence of restriction to perform physiotherapy | 24 hours
  Inability to perform physiotherapy secondary to pain or motor blockade
Incidence of restriction to perform physiotherapy | 48 hours
  Inability to perform physiotherapy secondary to pain or motor blockade
Postoperative plasmatic creatinine level | 48 hours
  Plasmatic creatinine level measured in mg/dL from a blood sample

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico Universidad de Chile, Santiago, Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
deidentified data under reasonable request

REFERENCES:
- [Background] Aso K, Izumi M, Sugimura N, Okanoue Y, Kamimoto Y, Yokoyama M, Ikeuchi M. Additional benefit of local infiltration of analgesia to femoral nerve block in total knee arthroplasty: double-blind randomized control study. Knee Surg Sports Traumatol Arthrosc. 2019 Jul;27(7):2368-2374. doi: 10.1007/s00167-018-5322-7. Epub 2018 Dec 8. PMID 30536047
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Bai JW, An D, Perlas A, Chan V. Adjuncts to local anesthetic wound infiltration for postoperative analgesia: a systematic review. Reg Anesth Pain Med. 2020 Aug;45(8):645-655. doi: 10.1136/rapm-2020-101593. Epub 2020 May 30. PMID 32474417
- [Background] Andersen LO, Kehlet H. Analgesic efficacy of local infiltration analgesia in hip and knee arthroplasty: a systematic review. Br J Anaesth. 2014 Sep;113(3):360-74. doi: 10.1093/bja/aeu155. Epub 2014 Jun 17. PMID 24939863
- [Background] Hubbard RC, Naumann TM, Traylor L, Dhadda S. Parecoxib sodium has opioid-sparing effects in patients undergoing total knee arthroplasty under spinal anaesthesia. Br J Anaesth. 2003 Feb;90(2):166-72. doi: 10.1093/bja/aeg038. PMID 12538372
- [Background] Harris SI, Kuss M, Hubbard RC, Goldstein JL. Upper gastrointestinal safety evaluation of parecoxib sodium, a new parenteral cyclooxygenase-2-specific inhibitor, compared with ketorolac, naproxen, and placebo. Clin Ther. 2001 Sep;23(9):1422-8. doi: 10.1016/s0149-2918(01)80117-x. PMID 11589257
- [Background] Stoltz RR, Harris SI, Kuss ME, LeComte D, Talwalker S, Dhadda S, Hubbard RC. Upper GI mucosal effects of parecoxib sodium in healthy elderly subjects. Am J Gastroenterol. 2002 Jan;97(1):65-71. doi: 10.1111/j.1572-0241.2002.05265.x. PMID 11808971
- [Background] Seangleulur A, Vanasbodeekul P, Prapaitrakool S, Worathongchai S, Anothaisintawee T, McEvoy M, Vendittoli PA, Attia J, Thakkinstian A. The efficacy of local infiltration analgesia in the early postoperative period after total knee arthroplasty: A systematic review and meta-analysis. Eur J Anaesthesiol. 2016 Nov;33(11):816-831. doi: 10.1097/EJA.0000000000000516. PMID 27428259
- [Background] Affas F, Eksborg S, Wretenberg P, Olofsson C, Stephanson N, Stiller CO. Plasma concentration of ketorolac after local infiltration analgesia in hip arthroplasty. Acta Anaesthesiol Scand. 2014 Oct;58(9):1140-5. doi: 10.1111/aas.12371. Epub 2014 Jul 31. PMID 25078268
- [Background] Laoruengthana A, Rattanaprichavej P, Reosanguanwong K, Chinwatanawongwan B, Chompoonutprapa P, Pongpirul K. A randomized controlled trial comparing the efficacies of ketorolac and parecoxib for early pain management after total knee arthroplasty. Knee. 2020 Dec;27(6):1708-1714. doi: 10.1016/j.knee.2020.10.005. Epub 2020 Nov 13. PMID 33197808
- [Background] Chan E, Howle R, Onwochei D, Desai N. Infiltration between the popliteal artery and the capsule of the knee (IPACK) block in knee surgery: a narrative review. Reg Anesth Pain Med. 2021 Sep;46(9):784-805. doi: 10.1136/rapm-2021-102681. Epub 2021 May 14. PMID 33990439
- [Background] Summers S, Mohile N, McNamara C, Osman B, Gebhard R, Hernandez VH. Analgesia in Total Knee Arthroplasty: Current Pain Control Modalities and Outcomes. J Bone Joint Surg Am. 2020 Apr 15;102(8):719-727. doi: 10.2106/JBJS.19.01035. No abstract available. PMID 31985507
- [Background] Sankineani SR, Reddy ARC, Eachempati KK, Jangale A, Gurava Reddy AV. Comparison of adductor canal block and IPACK block (interspace between the popliteal artery and the capsule of the posterior knee) with adductor canal block alone after total knee arthroplasty: a prospective control trial on pain and knee function in immediate postoperative period. Eur J Orthop Surg Traumatol. 2018 Oct;28(7):1391-1395. doi: 10.1007/s00590-018-2218-7. Epub 2018 May 2. PMID 29721648